CLINICAL TRIAL: NCT01805323
Title: A Retrospective Chart Review of OZURDEX® in Patients With Macular Edema
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMA-OZU-12-001
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Patients with macular edema previously treated with dexamethasone intravitreal implant (OZURDEX®) according to general clinical practice.
  Interventions: Drug: Dexamethasone Intravitreal Implant

INTERVENTIONS:
Drug: Dexamethasone Intravitreal Implant — Dexamethasone Intravitreal Implant (OZURDEX®) previously administered according to general clinical practice.
  Other Names: OZURDEX®

SUMMARY:
This retrospective chart review study will describe the history of patients with retinal disease with macular edema to whom OZURDEX® (dexamethasone intravitreal implant) is administered, and assess treatment patterns and visual outcomes. OZURDEX® was previously administered according to general clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Retinal disease involving macular edema
* Received at least one OZURDEX® injection

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with macular edema
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-04-15 (Actual); Study Completion 2013-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Québec, Quebec, Canada

REFERENCES:
- [Background] Lam WC, Albiani DA, Yoganathan P, Chen JC, Kherani A, Maberley DA, Oliver A, Rabinovitch T, Sheidow TG, Tourville E, Wittenberg LA, Sigouin C, Baptiste DC. Real-world assessment of intravitreal dexamethasone implant (0.7 mg) in patients with macular edema: the CHROME study. Clin Ophthalmol. 2015 Jul 10;9:1255-68. doi: 10.2147/OPTH.S80500. eCollection 2015. PMID 26203215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 66

OUTCOME MEASURES:

1. Primary Outcome: Peak Mean Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). The peak mean change in BCVA was calculated using the most improved number of lines read correctly between 2 and 26 weeks following the last available injection of OZURDEX® - the number of lines read correctly at Baseline. A positive change from Baseline indicated improvement.
Time Frame: Baseline, 2 to 26 weeks (wks) following last injection (up to 6.5 months)
Population: All participants with BCVA observations available following the last OZURDEX® injection from 2 to 26 weeks.
Measure: Mean (Standard Error); unit: Lines
Units Other Than Participants: Eyes
Arm/Group | All Participants
Number analyzed (Participants) | 78
Number analyzed (Eyes) | 90
Lines
  Baseline | 6.3 (0.3)
  Change from Baseline 2-26 wks after last injection | 1.4 (0.3)

2. Secondary Outcome: Peak Mean Change From Baseline in Central Retinal Thickness (CRT)
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye. The peak mean change was the maximum change from Baseline in CRT at 2 to 26 weeks following the last available injection of OZURDEX®. A negative change from Baseline indicated improvement.
Time Frame: Baseline, 2 to 26 weeks following last injection (up to 6.5 months)
Population: All participants with CRT observations available following the last OZURDEX® injection from 2 to 26 weeks.
Measure: Mean (Standard Error); unit: microns (μm)
Units Other Than Participants: Eyes
Arm/Group | All Participants
Number analyzed (Participants) | 75
Number analyzed (Eyes) | 85
microns (μm)
  Baseline | 474.4 (18.2)
  Change from Baseline 2-26 wks after last injection | -183.4 (17.9)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/101
Other Adverse Events (participants affected / at risk) | 25/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=101)
Endophthalmitis (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Retinal detachment (Injury, poisoning and procedural complications) | 1
Retinal implant (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=101)
Intraocular pressure increased (Investigations) | 19
Cystoid macular oedema (Eye disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.